CLINICAL TRIAL: NCT03644550
Title: Phase II Study of the Anti-Mesothelin Immunotoxin LMB-100 Followed by Pembrolizumab in Malignant Mesothelioma
Brief Title: Anti-Mesothelin Immunotoxin LMB-100 Followed by Pembrolizumab in Malignant Mesothelioma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to the Food and Drug Administration's recent approval of Nivolumab plus Ipilimumab as first line treatment for Mesothelioma, the principal investigator decided to end the study early (prior to reaching enrollment goal).
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Raffit Hassan, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 180136; 18-C-0136
Record Dates: First submitted 2018-08-22; First posted 2018-08-23 (Actual); Results first posted 2021-12-02 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Mesothelioma
Keywords: Checkpoint Inhibitor; Immunotherapy
MeSH Terms: conditions — Mesothelioma | interventions — LMB-100; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1/LMB- 100+pembrolizumab (Experimental): LMB-100 administered in cycles 1 and 2 + pembrolizumab administered in subsequent cycles.
  LMB-100 140mcg/kg Intravenous infusion (IVI), Days 1, 3, 5 in cycles 1, 2. Pembrolizumab 200mg IVI, every (Q) subsequent cycle on Day 1.
  Interventions: Drug: LMB-100; Biological: Pembrolizumab

INTERVENTIONS:
Drug: LMB-100 — Given intravenous (IV) at recommended phase 2 dose (RP2D) on days 1, 3 and 5 of two (2) 21 day cycles.
Biological: Pembrolizumab — Given intravenous (IV) at approved dose on day 1 of each 21 day cycle, starting with cycle 3, for up to 2 years with the option of a second course for patients meeting criteria.
  Other Names: Keytruda

SUMMARY:
Background:

Treatment outcomes for people with pleural or peritoneal mesothelioma are often poor. The drug LMB-100 can attack and kill cancer cells. The drug pembrolizumab helps the immune system fight cancer. Together, these drugs might help people with these cancers.

Objective:

To test if pembrolizumab given after LMB-100 shrinks tumors in people with pleural or peritoneal mesothelioma.

Eligibility:

People ages 18 and older with pleural or peritoneal mesothelioma that has not responded to platinum-based therapy

Design:

Participants will be screened with:

Tumor sample. Participants will have a biopsy if one is needed.

Medical history

Physical exam

Blood, heart, and urine tests

X-rays and scans: Participants will lie on a table. A machine will take pictures of the body.

Participants will receive LMB-100 by intravenous (IV) on days 1, 3, and 5 of two 21-day cycles. They will be observed for up to 2 hours after each infusion. They will receive drugs like Benadryl, Tylenol, and Zantac to help with side effects.

Starting with the 3rd cycle, participants will receive pembrolizumab by IV on day 1 of each 21-day cycle for up to 2 years.

Participants will have blood and urine tests, heart tests, and chest x-rays at least once per cycle. They will have scans every 6 weeks.

Participants may opt to provide tumor biopsies before starting the first cycle, after 2 cycles of LMB-100, and after 2 cycles of pembrolizumab.

Participants will a follow-up visit 4-6 weeks after their last drug dose of the study drug. This includes blood and heart tests and scans. They may then have scans every 6 weeks.

Participants will be contacted once a year for follow-up.

DETAILED DESCRIPTION:
Background:

* LMB-100, and a closely related immunotoxin, SS1P, also targeting mesothelin, have been studied in previous Phase 1 clinical studies for mesothelioma and pancreatic cancer.
* LMB-100 has demonstrated anti-tumor efficacy against several mesothelin expressing tumor models including mesothelioma patient-derived xenografts (PDX) models
* Programmed cell death protein 1 (PD-1) (encoded by the gene Pdcd1) is an Ig superfamily member related to cluster of differentiation 28 (CD28) and cytotoxic T lymphocyte-associated antigen-4 (CTLA-4) that has been shown to negatively regulate antigen receptor signaling upon engagement of its ligands
* The PD-1 receptor-ligand interaction is a major pathway hijacked by tumors to suppress immune control. The normal function of PD-1, expressed on the cell surface of activated T-cells under healthy conditions, is to down-modulate unwanted or excessive immune responses, including autoimmune reactions.
* In immune-competent mice bearing human mesothelin expressing tumors local administration of LMB-100 with CTLA-4 blockade eradicates murine tumors by promoting anti-cancer immunity.
* LMB-100 treatment increase cluster of differentiation 8 (CD8)+ T cell infiltration in murine lung adenocarcinoma tumors that express human mesothelin.
* Combination treatment with LMB-100 plus anti-PD1 results in greater anti-tumor efficacy in murine lung cancer model
* Pembrolizumab is an anti PD-1 antibody that has demonstrated responses of long duration in clinical trials and has generally been well-tolerated
* It is hypothesized that the anti-mesothelin immunotoxin LMB-100 followed by pembrolizumab will result in greater anti-tumor efficacy in patients with mesothelioma.

Objectives:

- To determine the objective response rate of sequential therapy with LMB-100 followed by pembrolizumab in subjects with pleural and peritoneal mesothelioma.

Eligibility:

* Histologically confirmed epithelial or biphasic pleural or peritoneal mesothelioma (with <50% sarcomatoid component) not amenable to potentially curative surgical resection.
* Subjects must have at least one prior chemotherapy regimen that includes pemetrexed and cisplatin or carboplatin.
* Age greater than or equal to 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate organ and bone marrow function
* Prior PD1/Programmed death-ligand 1 (PD-L1) inhibitor treatment is prohibited
* Chemotherapy within 4 weeks or radiotherapy within 2 weeks prior to start of study therapy is prohibited.
* Subjects with active central nervous system (CNS) metastasis are excluded
* Subjects with active autoimmune disease for which they had received systemic treatment during the previous 2 years receiving systemic glucocorticoids (excluding daily glucocorticoid-replacement therapy for conditions such as adrenal or pituitary insufficiency) are excluded
* Subjects with active interstitial lung disease, or a history of pneumonitis for which they had received glucocorticoids are excluded

Design:

* This is an open-label, single center phase II study of LMB-100 followed by pembrolizumab in subjects with advanced pleural or peritoneal mesothelioma who have progressed on standard therapies.
* Subjects will receive LMB-100 at the single agent maximum tolerated dose (MTD) on days 1, 3 and 5 of a 21-day cycle for 2 cycles and pembrolizumab 200 mg on day 1 of each subsequent 21-day cycle until disease progression (on or after pembrolizumab) or intolerable toxicity for a maximum of 2 years (unless second course initiated).
* Tumor biopsies will be performed at baseline, at the end of cycle 2 and at the end of cycle 4 to evaluate changes in the tumor immune microenvironment following treatment with LMB-100 and pembrolizumab.
* Up to 35 evaluable subjects will be enrolled

ELIGIBILITY:
* INCLUSION CRITERIA:

Participants are eligible to be included in the study only if all of the following criteria apply.

* Male and female participants who are at least 18 years of age on the day of signing the informed consent will be enrolled in the study.
* Subjects must have histologically confirmed diagnosis of:
* Cohort 1: Histologically confirmed epithelial or biphasic pleural mesothelioma (with <50% sarcomatoid component) not amenable to potentially curative surgical resection. The diagnosis will be confirmed by the Laboratory of Pathology, Center for Cancer Research (CCR), National Cancer Institute (NCI). OR
* Cohort 2: Histologically confirmed epithelial or biphasic peritoneal mesothelioma (with <50% sarcomatoid component) not amenable to potentially curative surgical resection. The diagnosis will be confirmed by the Laboratory of Pathology, CCR, NCI.
* Have provided archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides. Newly obtained biopsies are preferred to archived tissue.

Note: If submitting unstained cut slides, newly cut slides should be submitted to the testing laboratory within 14 days from the date slides are cut.

* Have measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Lesions in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
* Subjects must have at least one prior chemotherapy regimen that includes pemetrexed and cisplatin or carboplatin.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1. Evaluation of ECOG is to be performed within 7 days prior to start of study therapy.
* Have adequate organ and marrow function as defined below:

  * Hematological- hemoglobin: >= 9 g/dL or >= 5.6 mmol/L(a)
  * Hematological- absolute neutrophil count: >= 1,500/mcL
  * Hematological- platelets: >= 100,000/mcL
  * Hepatic- total bilirubin: less than or equal to 2.5 X institutional upper limit of normal (ULN) OR direct bilirubin less than or equal to ULN for participants with total bilirubin levels >1.5 X ULN
  * Hepatic- aspartate aminotransferase (AST) and alanine aminotransferase (ALT): less than or equal to 2.5 X institutional ULN (less than or equal to 5 X ULN for participants with liver metastases)
  * Renal-Creatinine less than or equal to 1.5 x ULN OR >= 50 mL/min for participant with creatinine levels > 1.5 X institutional ULN. Measured or calculated(b) creatinine clearance (Glomerular filtration rate (GFR) can also be used in place of creatinine or creatinine clearance (CrCl)
  * Coagulation-International normalized ratio (INR) OR prothrombin time (PT)/ Activated partial thromboplastin time (aPTT): less than or equal to 1.5 x ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants
  * ALT (SGPT)=alanine aminotransferase (serum glutamic pyruvic transaminase);
  * AST (SGOT)=aspartate aminotransferase (serum glutamic oxaloacetic transaminase);
  * GFR=glomerular filtration rate; ULN=upper limit of normal.
  * a. Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks.
  * b. Creatinine clearance (CrCl) or estimated glomerular filtration rate (eGFR) should be calculated per institutional standard.
* Must have left ventricular ejection fraction >50%.
* Must recovered from all adverse events (AEs) due to previous therapies to less than or equal to Grade 1 or baseline. Participants with less than or equal to Grade 2 neuropathy may be eligible. If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.
* Must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (less than or equal to 2 weeks of radiotherapy) to non-central nervous system (CNS) disease.
* If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.
* The effects of LMB-100 on the developing human fetus are unknown. For this reason and because anti-programmed cell death protein 1 (PD-1) antibodies such as pembrolizumab are assumed to be teratogenic:
* A male participant must agree to use contraception during the treatment period and for at least 180 days after the last dose of study treatment and refrain from donating sperm
* A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

  * Not a woman of childbearing potential (WOCBP) OR
  * A WOCBP who agrees to follow the contraceptive guidance in Appendix B during the treatment period and for at least 180 days after the last dose of study treatment.
* Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* The participant provides written informed consent for the trial.

EXCLUSION CRITERIA:

- Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.

Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.

* Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
* Has severe hypersensitivity (>= Grade 3) to pembrolizumab, LMB-100 and/or any of their excipients.
* Subjects who have received prior therapy with LMB-100, an anti-PD-1, anti-PD-L1, or anti-programmed cell death ligand 2 (PD-L2) agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., Cytotoxic T-lymphocyte antigen 4 (CTLA-4), OX-40, tumor necrosis factor receptor superfamily member 9 (CD137).
* Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to start of study therapy.
* Has received prior radiotherapy within 2 weeks of start of study treatment.
* Has had a prior pneumonectomy
* Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guerin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist(R)) are live attenuated vaccines and are not allowed.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to start of study therapy.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g.., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has a history of (non-infectious) pneumonitis/interstitial lung disease (ILD) that required steroids or has current pneumonitis/ILD
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* A WOCBP who has a positive urine pregnancy test within 72 hours prior to start of study therapy (see Appendix B). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. Note: in the event that 72 hours have elapsed between the screening pregnancy test and the first dose of study treatment, another pregnancy test (urine or serum) must be performed and must be negative in order for subject to start receiving study medication.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 180 days after the last dose of trial treatment. Pregnant women are excluded from this study because LMB-100 + pembrolizumab are agents with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with LMB-100 + pembrolizumab, breastfeeding should be discontinued if the mother is treated with LMB-100 + pembrolizumab. These potential risks may also apply to other agents used in this study.
* Has a known history of Human Immunodeficiency Virus. HIV positive patients will be excluded due to a theoretical concern that the degree of immune suppression associated with the treatment may result in progression of HIV infection. (Note: No HIV testing is required)
* Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV ribonucleic acid (RNA) [qualitative] is detected) infection. or active hepatitis B virus (HBV) or HCV infection. (Note: No testing for Hepatitis B and Hepatitis C is required.)
* Has a known additional malignancy that is progressing or has required active treatment within the past 2 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
* Has an active infection requiring systemic therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-12-04 (Actual); Primary Completion 2020-08-05 (Actual); Study Completion 2020-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raffit Hassan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2018-C-0136.html

RESULTS

PARTICIPANT FLOW:
Groups:
- 1/LMB- 100+Pembrolizumab: LMB-100 administered in cycles 1 and 2 + pembrolizumab administered in subsequent cycles.
  LMB-100 140mcg/kg Intravenous infusion (IVI), Days 1, 3, 5 in cycles 1, 2. Pembrolizumab 200mg IVI, every (Q) subsequent cycle on Day 1.
  LMB-100: Given intravenous (IV) at recommended phase 2 dose (RP2D) on days 1, 3 and 5 of two (2) 21 day cycles (i.e. RP2D was determined in a previous phase I trial).
  Pembrolizumab: Given intravenous (IV) at approved dose on day 1 of each 21 day cycle, starting with cycle 3, for up to 2 years with the option of a second course for patients meeting criteria.
Period: Overall Study
Arm/Group | 1/LMB- 100+Pembrolizumab
Started | 18
Completed | 0
Not Completed | 18
Not completed — Withdrawal by Subject | 3
Not completed — Progressive disease | 15

BASELINE CHARACTERISTICS:
Groups:
- 1/LMB- 100+Pembrolizumab: LMB-100 administered in cycles 1 and 2 + pembrolizumab administered in subsequent cycles.
  LMB-100 140mcg/kg Intravenous infusion (IVI), Days 1, 3, 5 in cycles 1, 2. Pembrolizumab 200mg IVI, every (Q) subsequent cycle on Day 1.
  LMB-100: Given intravenous (IV) at recommended phase 2 dose (RP2D) on days 1, 3 and 5 of two (2) 21 day cycles (i.e. RP2D was determined in a previous phase I trial)..
  Pembrolizumab: Given intravenous (IV) at approved dose on day 1 of each 21 day cycle, starting with cycle 3, for up to 2 years with the option of a second course for patients meeting criteria.
Arm/Group | 1/LMB- 100+Pembrolizumab
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.62 (12.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Objective Response (Partial Response + Complete Response)
Description: Number of participants who received at least 1 cycle of study therapy and who had their disease reevaluated that experienced a partial or complete response per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 or modified RECIST criteria. Complete Response is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: Every 6 weeks until disease progression, an average of 3.1 months
Population: 17/18 participants were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | 1/LMB- 100+Pembrolizumab
Number analyzed (Participants) | 17
Participants
  Partial Response | 3
  Complete Response | 0

2. Secondary Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0).
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 22 months and 29 days.
Measure: Count of Participants; unit: Participants
Arm/Group | 1/LMB- 100+Pembrolizumab
Number analyzed (Participants) | 18
Participants | 18

3. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression free survival (PFS) is defined as the duration of time from start of treatment to time of progression (on or after pembrolizumab) or death, whichever occurs first. Progression was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST). Progression is at least a 20% increase in the sum of the diameters of target lesions,taking as reference the smallest sum on study.
Time Frame: Time from start of treatment to time of progression (on or after pembrolizumab) or death, whichever occurs first, an average of 6.5 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 1/LMB- 100+Pembrolizumab
Number analyzed (Participants) | 18
Months | 7.1 [4.3 to 8.4]

4. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is the time between the first day of treatment to the day of death.
Time Frame: Time between the first day of treatment to the day of death, an average of 17 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 1/LMB- 100+Pembrolizumab
Number analyzed (Participants) | 18
Months | 17.1 [10.2 to 27.5]

5. Secondary Outcome: Duration of Overall Response (DOR)
Description: The duration of overall response is measured from the time measurement criteria are met for complete response (CR) or partial response (PR) (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented. Response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST). Complete Response (CR) is defined as disappearance of all target lesions with no evidence of tumor elsewhere. Partial Response (PR) is defined as at least a 30% decrease in the total tumor measurement.
Time Frame: Time measurement criteria are met for complete response (CR) or partial response (PR) (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented, an average of 3.1 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 1/LMB- 100+Pembrolizumab
Number analyzed (Participants) | 18
Months | 3.1 [2.8 to 11.7]

6. Secondary Outcome: Percentage of Participants With an Overall Response
Description: Percentage of participants who received at least 1 cycle of study therapy and who had their disease reevaluated that experienced a partial or complete response per the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 or modified RECIST criteria. Complete Response is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: An average of 3.1 months.
Population: 17/18 participants were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | 1/LMB- 100+Pembrolizumab
Number analyzed (Participants) | 17
percentage of participants | 17.6

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 22 months and 29 days.
Arm/Group | 1/LMB- 100+Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 9/18
Serious Adverse Events (participants affected / at risk) | 14/18
Other Adverse Events (participants affected / at risk) | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1/LMB- 100+Pembrolizumab (N=18)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 3 (4)
CPK increased (Investigations) | 1 (1)
Capillary leak syndrome (Vascular disorders) | 2 (2)
Colitis (Gastrointestinal disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Small intestinal perforation (Gastrointestinal disorders) | 1 (2)
Thyroid stimulating hormone increased (Investigations) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1/LMB- 100+Pembrolizumab (N=18)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 7 (9)
Activated partial thromboplastin time prolonged (Investigations) | 7 (14)
Alanine aminotransferase increased (Investigations) | 14 (21)
Alkaline phosphatase increased (Investigations) | 6 (14)
Anemia (Blood and lymphatic system disorders) | 17 (109)
Anorexia (Metabolism and nutrition disorders) | 7 (9)
Anxiety (Psychiatric disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 13 (24)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (7)
Bacteremia (Infections and infestations) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 2 (2)
CPK increased (Investigations) | 2 (4)
Capillary leak syndrome (Vascular disorders) | 1 (1)
Cardiac troponin I increased (Investigations) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (14)
Creatinine increased (Investigations) | 13 (32)
Depression (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 6 (6)
Dizziness (Nervous system disorders) | 6 (9)
Dry eye (Eye disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Dysgeusia (Nervous system disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 3 (5)
Dysphagia (Gastrointestinal disorders) | 2 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Edema face (General disorders) | 1 (1)
Edema limbs (General disorders) | 3 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (2)
External ear pain (Ear and labyrinth disorders) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Fatigue (General disorders) | 10 (18)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Fever (General disorders) | 4 (6)
Flank pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Floaters (Eye disorders) | 1 (1)
Flushing (Vascular disorders) | 2 (2)
Folliculitis (Infections and infestations) | 1 (1)
GGT increased (Investigations) | 1 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, Abdominal pain (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, Alveolar bone loss (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, Left side jaw pain (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, Wisdom tooth extraction (Gastrointestinal disorders) | 2 (4)
Generalized edema (General disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 9 (17)
Hematuria (Renal and urinary disorders) | 2 (2)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 3 (9)
Hyperglycemia (Metabolism and nutrition disorders) | 8 (38)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 (4)
Hyperkalemia (Metabolism and nutrition disorders) | 6 (10)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (3)
Hypernatremia (Metabolism and nutrition disorders) | 2 (3)
Hyperphosphatemia (Metabolism and nutrition disorders) | 4 (6)
Hypertension (Vascular disorders) | 6 (17)
Hyperthyroidism (Endocrine disorders) | 2 (2)
Hyperuricemia (Metabolism and nutrition disorders) | 3 (5)
Hypoalbuminemia (Metabolism and nutrition disorders) | 16 (55)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (5)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 4 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 5 (9)
Hyponatremia (Metabolism and nutrition disorders) | 10 (33)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (6)
Hypotension (Vascular disorders) | 8 (10)
Hypothyroidism (Endocrine disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 3 (3)
Insomnia (Psychiatric disorders) | 4 (5)
Investigations - Other, RBC Urin increased (Investigations) | 1 (1)
Investigations - Other, WBC Urine (Investigations) | 1 (3)
Investigations - Other, pro Brain Natriuretic peptide (Investigations) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1)
Localized edema (General disorders) | 10 (19)
Lung infection (Infections and infestations) | 1 (1)
Lymphocyte count decreased (Investigations) | 17 (74)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 9 (18)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — - Other, Melanoma (noted lesion 4 months ago on right upper arm)
Neutrophil count decreased (Investigations) | 2 (6)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 5 (9)
Oral pain (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 5 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (9)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Papulopustular rash (Skin and subcutaneous tissue disorders) | 2 (2)
Paresthesia (Nervous system disorders) | 1 (4)
Penile infection (Infections and infestations) | 1 (1)
Pericardial effusion (Cardiac disorders) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Platelet count decreased (Investigations) | 5 (9)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Presyncope (Nervous system disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 3 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (4)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Sinus tachycardia (Cardiac disorders) | 8 (12)
Skin and subcutaneous tissue disorders - Other, Erythema abigne (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 1 (1) — - Other, Keratosis ( right forearm, left forehead, right eyebrow
Skin and subcutaneous tissue disorders - Other,Left arm distal to IV site (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Lesion right forearm (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, left shoulder and left leg (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, pimple located on top of gluteal cleft (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Syncope (Nervous system disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Thyroid stimulating hormone increased (Endocrine disorders) | 5 (8)
Toothache (Gastrointestinal disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (7)
Weight gain (Investigations) | 10 (16)
Weight loss (Investigations) | 7 (13)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
White blood cell decreased (Investigations) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-16): https://cdn.clinicaltrials.gov/large-docs/50/NCT03644550/Prot_SAP_000.pdf
  • Informed Consent Form (2020-09-15): https://cdn.clinicaltrials.gov/large-docs/50/NCT03644550/ICF_001.pdf